CLINICAL TRIAL: NCT05767983
Title: Effect of Dairy on Cognitive Performance, Subjective Appetite and Glycemic Response in Children
Brief Title: Effect of Dairy on Cognitive Performance in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Dairy Management Inc. (Industry); National Dairy Council (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, PhD, Associate Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Temp ID
Record Dates: First submitted 2022-11-23; First posted 2023-03-14 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Children; Healthy
Keywords: Cognitive performance; Appetite; Mood; Glycemic response; Emotions; Dairy consumption
MeSH Terms: interventions — Fruit and Vegetable Juices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Fat-free milk (Experimental): Treatment
  Interventions: Other: Fat-free milk
- Fat-free yogurt (Experimental): Treatment
  Interventions: Other: Fat-free yogurt
- Low-fat cheese (Experimental): Treatment
  Interventions: Other: Low-fat cheese
- Fruit juice (Experimental): Treatment
  Interventions: Other: Fruit juice
- Snack skipping (Experimental): Treatment
  Interventions: Other: Snack skipping

INTERVENTIONS:
Other: Fat-free milk — Fat-free milk (500 mL, skim, 0%, Lactantia PurFiltre) will provide 180 kcal, 0 g fat, 26 g carbohydrate, and 18 g protein. Treatments matched for calories (180 kcal).
  Arms: Fat-free milk
Other: Fat-free yogurt — Fat-free yogurt (242 g, vanilla, 0% Greek, Oikos) will provide 180 kcal, 0 g fat, 23.5 g carbohydrate, and 19.4 g protein. Treatments matched for calories (180 kcal).
  Arms: Fat-free yogurt
Other: Low-fat cheese — Low-fat cheese (60 g, mild marble cheddar, 40% less fat, Selection) will provide 180 kcal, 10 g fat, 2 g carbohydrate, and 16 g protein. Treatments matched for calories (180 kcal).
  Arms: Low-fat cheese
Other: Fruit juice — Fruit juice (450 mL, Fruité® Fruit Punch) will provide 180 kcal, 0 g fat, 46.8 g carbohydrate, and 0 g protein. Treatments matched for calories (180 kcal).
  Arms: Fruit juice
Other: Snack skipping — Water control treatment (no caloric contribution). Matched for volume (500 mL) to fat-free milk treatment.
  Arms: Snack skipping

SUMMARY:
The purpose of this study is to determine the effects of dairy consumption on short-term cognitive performance, subjective mood and emotions, and glycemic response in healthy children aged 9 - 14 years. The investigators hypothesize that the consumption of dairy products as a mid-morning snack will improve mood and cognitive performance in children. Furthermore, the investigators hypothesize that all dairy products consumed as a mid-morning snack will imbue more benefits on mood and cognitive performance over 2-hours compared to fruit juice or snack skipping.

DETAILED DESCRIPTION:
A randomized within-subject repeated measures experiment will be used to study the effects of dairy product consumption on cognitive performance, subjective mood and emotions, and blood glucose in healthy 9 - 14 year old children. Participants will consume, in a random order on separate mornings, one of the five treatments: (a) milk, (b) yogurt, (c) cheese, (d) fruit juice, or (e) snack skipping. Subjective mood/emotions and cognitive domains (learning and memory, spatial working memory, attention, processing speed, and executive function) will be assessed at baseline (0-min), and 15-, 30-, 60-, and 120-min following treatment consumption. Blood glucose measurements will be collected using the Freestyle Libre 2 continuous glucose monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* 9 to 14 years of age;
* Normal weight defined as between the 15th and 80th percentile for age and biological sex at birth according to the World Health Organization growth (WHO) charts.

Exclusion Criteria:

* Children with overweight/ obesity;
* Children with food sensitivities or allergies to dairy, gluten or any foods used in the study;
* Children with any diagnosed learning, emotional, or behavioural disabilities;
* Children taking any medications that may influence cognitive performance.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Learning and short-term memory | Change from baseline (measured at 0-minutes before treatment) and at 15-minutes, 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Learning and short-term memory will be assessed using an immediate and delayed Word Recall Test (accuracy).
Spatial working memory | Change from baseline (measured at 0-minutes before treatment) and at 15-minutes, 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Spatial working memory will be assessed using the forward and backward versions of the Corsi Block Test (accuracy).
Sustained attention | Change from baseline (measured at 0-minutes before treatment) and at 15-minutes, 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Sustained attention and processing speed will be assessed using the Continuous Performance Test (CPT) (accuracy and reaction time).
Executive function | Change from baseline (measured at 0-minutes before treatment) and at 15-minutes, 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  Cognitive performance tests will be administered via a Dell tablet (Millisecond, Inquisit Web) and paper/pen. Executive function and selective attention will be assessed using the Flanker Task (accuracy and reaction time).

SECONDARY OUTCOMES:
Glycemic response | Change from baseline (measured at 0-minutes before treatment) and 15-minutes, 30-minutes, 45-minutes, 60-minutes, 75-minutes, 90-minutes, 105-minutes and 120-minutes post-treatment consumption
  Blood glucose (mmol/L). Blood glucose concentrations will be measured using a Freestyle Libre 2 continuous glucose monitoring (CGM) and flash-glucose system.
Subjective mood and emotion | Change from baseline (measured at 0-minutes before treatment) and at 15-minutes, 30-minutes, 60-minutes and 120-minutes post-treatment consumption
  A visual analogue scale (VAS) with thirteen questions will be administered to assess subjective emotions and mood (aggression, anger, excitement, disappointment, happiness, upset, frustration, alertness, sadness, tension, exhaustion, calmness, sleepiness, and wellness). Individual questions will be used to form a composite emotion score. Each VAS will be administered via a digital software application (Express VAS, Toronto, Ontario, Canada) on a Dell tablet where children will place an 'X" on the VAS line (100 unit scale) to describe their feelings.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PhD, Principal Investigator — Toronto Metropolitan University
Locations (1):
- Centre for Urban Innovation (CUI-109), Toronto Metropolitan University (Formerly Ryerson University), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No